CLINICAL TRIAL: NCT06861946
Title: Silicone Effect on Corneal Endothelium and Corneal Biomechanics Using Corvis ST
Status: Completed | Type: Observational
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mohamed Yasser Sayed Saif, Dean of National Institute of Longvity Elder Sciences, Beni-Suef University
Other Study IDs: R241/R242
Record Dates: First submitted 2025-02-21; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Silicon Oil Effect on Cornea; Corneal Biomechanics
Keywords: Corneal biomechanics; Specular microscopy; silicon oil; endothelial cell density

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Group (A): Vitrectomy with 1000 cSt silicone oil.
  Interventions: Diagnostic Test: Corvis ST; Diagnostic Test: Conrneal endothelial cell density
- group (B): Phaco vitrectomy with 1000 cSt silicone oil.
  Interventions: Diagnostic Test: Corvis ST; Diagnostic Test: Conrneal endothelial cell density
- group (C): Vitrectomy with 5000 cSt silicone oil.
  Interventions: Diagnostic Test: Corvis ST; Diagnostic Test: Conrneal endothelial cell density
- group (D): Phaco vitrectomy with 5000 cSt silicone oil.
  Interventions: Diagnostic Test: Corvis ST; Diagnostic Test: Conrneal endothelial cell density
- group (E): Control group (other eyes).
  Interventions: Diagnostic Test: Corvis ST; Diagnostic Test: Conrneal endothelial cell density

INTERVENTIONS:
Diagnostic Test: Corvis ST — Corvis ST is used to assess corneal biomechanical changes following vitrectomy with silicone oil tamponade, specifically:
  Corneal stiffness and elasticity using the Stress-Strain Index (SSI) Corneal deformation response via Deformation Amplitude (DA)
  Other Names: Corneal Biomechanics
Diagnostic Test: Conrneal endothelial cell density — The study evaluates the impact of silicone oil tamponade on corneal endothelial cell density (ECD) in patients undergoing vitrectomy for retinal detachment. The intervention involves:
  Preoperative and Postoperative Assessments at 1, 3, and 6 months to monitor changes in ECD.
  Specular Microscopy to measure ECD (cells/mm²), coefficient of variation (CV) in cell size, and hexagonality (% of hexagonal cells).

SUMMARY:
Brief Summary

The goal of this observational study is to investigate the effects of silicone oil tamponade on corneal endothelial cell density (ECD), morphology, and biomechanics in patients undergoing vitrectomy for retinal detachment (20 patients, 20 eyes). The main questions it aims to answer are:

How does silicone oil tamponade affect corneal ECD, morphology, and biomechanics over 6 months postoperatively?

Are these changes associated with variations in best-corrected visual acuity (BCVA) or intraocular pressure (IOP)?

Comparison group: Researchers will compare preoperative measurements to 1-, 3-, and 6-month postoperative assessments to evaluate changes in endothelial parameters and corneal biomechanics.

Participants will:

Undergo preoperative and postoperative assessments (at 1, 3, and 6 months) using specular microscopy (to measure ECD, coefficient of variation, hexagonality) and Corvis ST (to evaluate biomechanical properties: Stress-Strain Index and deformation amplitude).

Have BCVA and IOP measured at each follow-up visit to track clinical outcomes.

DETAILED DESCRIPTION:
This prospective observational study evaluates the impact of silicone oil tamponade on corneal endothelial integrity and biomechanical properties in patients undergoing vitrectomy for retinal detachment. Below is an expanded description of the study protocol, emphasizing methodological rigor and technical specifics.

Study Design Type: Single-center, prospective, longitudinal observational study. Primary Objective: To quantify postoperative changes in corneal endothelial cell density (ECD), morphology, and biomechanical stability over a 6-month period following silicone oil tamponade.

Secondary Objectives:

Correlate corneal changes with clinical outcomes (BCVA, IOP).

Identify risk factors for endothelial cell loss or biomechanical weakening.

Rationale for Time Points: Assessments at 1, 3, and 6 months were selected to capture early postoperative stress responses (1 month), intermediate healing (3 months), and longer-term stabilization (6 months), aligning with standard vitrectomy follow-up protocols.

Participant Enrollment Recruitment: Consecutive patients scheduled for vitrectomy with silicone oil tamponade at a tertiary eye care center.

Informed Consent Process: Participants received detailed verbal and written explanations of study procedures, risks, and benefits prior to enrollment.

Data Collection Procedures Clinical and Imaging Assessments

Best-Corrected Visual Acuity (BCVA):

Measured using Snellen charts under standardized lighting conditions.

Converted to logMAR for statistical analysis.

Intraocular Pressure (IOP):

Assessed via Goldmann applanation tonometry (calibrated weekly), with three consecutive readings averaged.

Corneal Endothelial Analysis:

Specular Microscopy (Konan Noncon Robo NSP-9900):

Parameters:

Endothelial Cell Density (ECD): Cells/mm².

Coefficient of Variation (CV): Reflects cell size variability (polymegathism).

Hexagonality: Percentage of hexagonal cells (pleomorphism).

Protocol: Central corneal measurements taken in triplicate, with the median value recorded.

Corneal Biomechanical Evaluation:

Corvis ST (Oculus Optikgeräte GmbH):

Parameters:

Stress-Strain Index (SSI): Quantifies corneal stiffness.

Deformation Amplitude (DA): Maximum corneal displacement during air-puff applanation.

Protocol: Three valid scans per eye, performed under mesopic conditions.

Follow-Up Protocol Baseline: Preoperative assessment within 1 week of surgery.

Postoperative: Follow-up visits at 1, 3, and 6 months (±7 days), including:

BCVA and IOP measurement.

Specular microscopy and Corvis ST imaging.

Documentation of complications (e.g., corneal edema, elevated IOP).

Quality Assurance Measures

Equipment Calibration:

Specular microscopy and Corvis ST devices underwent daily calibration checks and quarterly manufacturer servicing.

Standardized Protocols:

All measurements performed by a single trained ophthalmologist to minimize inter-observer variability.

Consistent time-of-day scheduling for IOP assessments (9 AM-11 AM) to control diurnal fluctuations.

Blinded Analysis:

Endothelial and biomechanical data were analyzed by masked investigators unaware of clinical outcomes or time points.

Data Management and Statistical Analysis

Data Storage:

Clinical and imaging data stored in a HIPAA-compliant REDCap database with role-based access.

Regular backups to encrypted cloud storage.

Statistical Methods:

Primary Analysis: Linear mixed-effects models to evaluate longitudinal changes in ECD, SSI, and DA.

Secondary Analysis: Pearson/Spearman correlations between endothelial parameters, biomechanics, and BCVA/IOP.

Missing Data: Multiple imputation used for sporadic missing follow-up data (<10% attrition anticipated).

Software: Analyses performed using R (v4.3.1) and SPSS (v28.0).

Ethical and Safety Considerations

Adverse Event Management:

Complications (e.g., corneal decompensation, IOP spikes) were managed per institutional guidelines and reported to the IRB.

Protocol Compliance:

Internal audits conducted quarterly to ensure adherence to GCP and study protocols.

Technical Rationale Silicone Oil Tamponade: While effective for retinal reattachment, silicone oil may mechanically stress the corneal endothelium or alter aqueous humor dynamics, potentially accelerating cell loss.

Biomechanical Relevance: Corneal stiffness (SSI) and deformability (DA) are critical for refractive stability and surgical planning (e.g., cataract surgery post-vitrectomy).

Clinical Implications

This study aims to provide evidence-based recommendations for:

Timing of silicone oil removal to mitigate corneal damage.

Enhanced monitoring strategies for high-risk patients.

Personalized interventions to preserve endothelial health.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing vitrectomy.
* Clear cornea.
* Central corneal thickness (CCT) ≥ 500 µm.
* Age between 20 and 50 years.

Exclusion Criteria:

* History of intraocular surgery.
* Ocular pathologies, such as corneal scarring or dystrophy.
* Advanced keratoconus.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients undergoing vitrectomy with silicone oil tamponade for the treatment of rhegmatogenous retinal detachment (RRD).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Corneal Endothelial Cell Density (ECD) | Baseline (preoperative), 1 month, 3 months, and 6 months postoperatively.
  Measurement: Cells/mm², assessed via specular microscopy (Konan Noncon Robo NSP-9900).
Morphological Changes in Corneal Endothelium | Baseline, 1, 3, and 6 months.
  Parameters:
  Coefficient of Variation (CV): Reflects cell size variability (polymegathism).
  Hexagonality: Percentage of hexagonal cells (pleomorphism).
  Measurement: Specular microscopy.
  CV and hexagonality are vital for evaluating corneal endothelial health. Optimal outcomes are associated with low CV (<30%) and high hexagonality (>60%), while deviations signal pathology or risk. Specular microscopy remains the gold standard for non-invasive assessment.
Corneal Biomechanical Properties | Baseline, 1, 3, and 6 months.
  Parameters:
  Stress-Strain Index (SSI): Quantifies corneal stiffness.
  Deformation Amplitude (DA): Maximum corneal displacement during air-puff applanation.
  Measurement: Corvis ST (Oculus Optikgeräte GmbH).
  Normal Ranges:
  SSI: Typically ranges between ~50-100 (unitless), though values vary by population and device software.
  DA: Normal corneas average ~1.0-1.2 mm, while keratoconic corneas often exceed 1.3 mm.

SECONDARY OUTCOMES:
Best-Corrected Visual Acuity (BCVA) | Baseline, 1, 3, and 6 months.
  Snellen charts converted to logMAR for analysis.
Intraocular Pressure (IOP) | Baseline, 1, 3, and 6 months.
  Goldmann applanation tonometry (average of three readings).
Correlation Between Corneal Changes and Clinical Outcomes | Baseline, 1, 3, and 6 months.
  Associations between ECD, biomechanical parameters (SSI/DA), and BCVA/IOP using regression models.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Fayoum University Hospital, Al Fayyum, Faiyum Governorate
  - Misr University For Science and Technology, Giza

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Goezinne F, Nuijts RM, Liem AT, Lundqvist IJ, Berendschot TJ, Cals DW, Hendrikse F, La Heij EC. Corneal endothelial cell density after vitrectomy with silicone oil for complex retinal detachments. Retina. 2014 Feb;34(2):228-36. doi: 10.1097/IAE.0b013e3182979b88. PMID 23807185
- [Background] Latkowska M, Gajdzis M, Kaczmarek R. Emulsification of Silicone Oils: Altering Factors and Possible Complications-A Narrative Review. J Clin Med. 2024 Apr 20;13(8):2407. doi: 10.3390/jcm13082407. PMID 38673681